CLINICAL TRIAL: NCT01146444
Title: Investigation of the Efficacy of Different Sunscreens in Patients With Photosensitive Cutaneous Lupus Erythematosus
Brief Title: Sunscreens in Patients With Cutaneous Lupus Erythematosus(CLE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spirig Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DL0814-SPRG0801/KHMR
Record Dates: First submitted 2010-05-24; First posted 2010-06-17 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2013-12

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: Sunscreening Agents
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sunscreens with a low, medium, high SPF (Experimental): sunscreens with a low, medium, and high SPF. UVA and UVB irradiation
  Interventions: Other: UV A and B irradiation
- vehicle (Experimental): Intra-individual application of vehicle in random order; UVA and UVB irradiation
  Interventions: Other: UV A and B irradiation

INTERVENTIONS:
Other: UV A and B irradiation — UV irradiation

SUMMARY:
Part I: to investigate the efficacy of different sunscreens in the prevention of skin lesions following standardized photoprovocation with Ultraviolet A/Ultraviolet B (UVA/UVB) light in patients with CLE.

Part II: to evaluate the influence of different sunscreens on the expression of biomarkers in the skin of patients with CLE and of Healthy Controls following UV irradiation.

DETAILED DESCRIPTION:
Part I

Part I-interventions will be:

* Experimental intervention: Application of broad-spectrum sunscreens with a low, medium, and high Sun Protection Factor (SPF) in random order to uninvolved skin areas prior to standardized photoprovocation.
* Control intervention: Intra-individual application of vehicle in random order; standardized photoprovocation of vehicle treated and untreated areas.

Part II

Part II-interventions will be:

* Experimental intervention: Application of a broad-spectrum sunscreen with a high SPF to uninvolved skin areas prior to UV irradiation.
* Control intervention: UV irradiation of untreated areas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subacute cutaneous lupus erythematosus (SCLE), discoid lupus erythematosus (DLE), or lupus erythematosus tumidus (LET) according to the Düsseldorf Classification 2004 (Kuhn and Ruzicka 2004) confirmed by histological analysis.
* Women of childbearing potential with a negative pregnancy test at screening (urine test) and using a medically accepted contraceptive regimen (intra-uterine device, partner's vasectomy, >3 months previous hormonal contraception (oestrogen plus gestagen pill, depot injections, or subcutaneous depot) combined with a barrier method (preservative, vaginal diaphragm, cervical cap, spermicide) during the study and for 8 weeks after the last UV exposure.
* Women clinically sterile (post-menopausal, undergone hysterectomy or tubal ligation).
* Actively cooperating to participate in the study, to follow the instructions of the investigator and to attend the centre at the agreed times.
* Development of skin lesions any time under current systemic treatment if patient is receiving systemic medication for the treatment of CLE.
* Signed informed consent form after the nature of the study has been fully explained.

Exclusion Criteria:

* Pregnancy or lactation and women with positive pregnancy test.
* Known hypersensitivity or allergic contact reactions to components of the study agents.
* Treatment with photosensitizing drugs.
* Exposure to direct natural (sunlight) or artificial UV radiation on the back within 4 weeks prior to entering the study.
* History of another photodermatosis, except polymorph light eruption (PLE).
* Any current known skin malignancy or any history of skin malignancy within the previous 5 years or Xeroderma pigmentosum.
* Initiation or change in the dose of any current systemic medication for the treatment of CLE within 8 weeks prior to standardized photoprovocation.
* Local therapy for the treatment of CLE within two weeks prior to standardized photoprovocation at the back of the patient
* Acute exacerbation of CLE skin disease within 2 weeks prior to entering the study.
* Acute illness within 7 days prior to phototesting or major illness including infection or hospitalization within 1 month of study entry.
* Anti-dsDNA (RIA) > 7 U/ml and/or at least one of the following criteria:
* Serositis: pleuritis or pericarditis documented by electrocardiogram or rub or evidence of pericardial effusion;
* Renal disorder: proteinuria greater than 0.5 g/d or greater than 3+, or cellular casts;
* Neurologic disorder: seizures or psychosis without other cause.
* Patients with a documented HIV and/or hepatitis B or C infection.
* Any medical condition, which would place the subject at undue risk of, or make it unlikely that follow-up-measurements could be obtained

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Prevention of skin lesions following standardized photoprovokation with UVA/UVB light in patients with CLE | September 2011

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Kuhn, MD, Principal Investigator — Professor
Locations (1):
- Klinik und Poliklinik für Hautkrankheiten, Universitätsklinikum Münster, Münster, Germany